CLINICAL TRIAL: NCT02202655
Title: Study of Changes of Lymphocyte Subsets in Chemotherapy Course of Patients With Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Yingmin Ma, Vice President of the Beijing chaoyang hospital, Beijing Chao Yang Hospital
Other Study IDs: 13501185982
Record Dates: First submitted 2014-06-24; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non- small cell lung cancer;; lymphocyte subsets
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the changes of lymphocyte subsets in chemotherapy course of patients with non-small cell lung cancer

DETAILED DESCRIPTION:
patients with primary non-small cell lung cancer who received first chemotherapy in Beijing Chaoyang Hospital affiliated to Capital Medical University were collected, and the percentage of lymphocyte subsets at 9 time points before, during, and after chemotherapy was detected by flow cytometry method.We will investigate the changes of patients' lymphocyte subsets in chemotherapy courses. The correlation of the percentage of lymphocyte subsets and age, gender, pathological type, clinical stage, surgery or not, clinical efficacy assessment will be further analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Each Period Non-small Cell Lung Cancer, Which Was Confirmed by Histopathology. patients has only lung cancer .
* Functional Status Score (PS) ≧ 70.
* The first time for chemotherapy .
* A Written Informed Consent.

Exclusion Criteria:

* Merging other tumors.
* HAve autoimmune diseases.
* AIDS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with non-small cell lung cancer who accept chemotherapy for the first time are acceptable.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
the changes of patients' lymphocyte subsets in chemotherapy courses. | up to cycle 4 day 9

CONTACTS AND LOCATIONS:
Overall Officials: yingmin ma, Study Director — Vice President of the Beijing chaoyang hospital
Locations (1):
- WangQian, Beijing, Beijing Municipality, China